CLINICAL TRIAL: NCT05113914
Title: The Influence of Age and Physical Fitness Level on the Level of Energy Metabolism and Antioxidant Capacity in Adult Males
Brief Title: The Age-related Changes of Energy Metabolism in Physically Fit Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: AWF_LA_MA865862
Record Dates: First submitted 2021-10-07; First posted 2021-11-09 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-09

CONDITIONS: Healthy
Keywords: athletes; masters; purine metabolites; NAD metabolites; CPET

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy, physically fit men (Experimental): All participants underwent a single CPET test with pre- and post-exercise blood measurements.
  Interventions: Diagnostic Test: Cardio-pulmonary exercise test

INTERVENTIONS:
Diagnostic Test: Cardio-pulmonary exercise test — An incremental running test was conducted on the treadmill. Initially, the exercise protocol included standing still for 3 min and walking for 3 min at a constant speed of 4 km/h. After this introductory part, the speed was increased to 8 km/h and then every 3 min by 2 km/h until the volitional exhaustion was reached. During all procedure oxygen consumption was measured with the use of a portable breath-by-breath ergospirometer.

SUMMARY:
The influence of age and physical fitness level on the level of energy metabolism and antioxidant capacity in adult males.

DETAILED DESCRIPTION:
Over four hundred healthy, adult males of different age categories and physical fitness levels were included in the study. There is much research convincing that in athletes of various sports disciplines the level of energy metabolism, oxidative stress, and amino acid profiles during years of training undergoes sports adaptation. The study aimed to evaluate how age and physical fitness level affects the level of purine metabolites and metabolites of nicotinamide adenine dinucleotide, the level of antioxidant capacity, and amino acid profiles. Investigators hypothesized that there will be an age-related decline in most of the physiological indices, but significant differences will appear regarding the level of an individual's sports adaptation.

ELIGIBILITY:
Inclusion Criteria:

1. healthy
2. non-smoking
3. physically fit, including top-level athletes

Exclusion Criteria:

1. no reported history of a cardiopulmonary or renal diseases, and other chronic diseases
2. no major orthopedic injury or illness resulting in an inability to run
3. no medications that could affect cardiopulmonary functions
4. normal resting electrocardiogram
5. body mass index (BMI) below 30.0 kg·m-2
6. normal erythrocyte count and Hb content
7. no pathological states known of significantly elevated adenylate pool and concentration of ATP, e.g. sickle cell disease, diabetes, leukemia, sepsis, tuberculosis, meningococcal infection, or renal insufficiency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only males were included in the study.
Enrollment: 420 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Cardio-respiratory measures | during the intervention
  Cardiopulmonary exercise test (CPET) was conducted while an incremental running test on the treadmill using a portable breath-by-breath ergospirometer and heart rate monitor.

SECONDARY OUTCOMES:
Blood Lactate level | baseline and immediately after the intervention
  Lactate concentration was performed by the spectrophotometric enzymatic method.
Plasma purine nucleotides | baseline and immediately after the intervention
  The plasma purine metabolites were estimated in plasma using high-performance liquid chromatography (HPLC) with UV-VIS detection.
  Measurements performed: Guanosine, Inosine, Adenosine, Hypoxanthine, Xanthine, Uric Acid, Allantoin, Adenine Nucleotides [adenosine triphosphate (ATP), adenosine diphosphate (ADP), adenosine monophosphate (AMP), inosine monophasphate (IMP)], Guanine Nucleotides [guanosine triphosphate (GTP), guanosine diphosphate (GDP), guanosine monophosphate (GMP)].
Erythrocyte Purine Metabolites | baseline and immediately after the intervention
  The erythrocyte purine metabolites were estimated in erythrocytes using high-performance liquid chromatography (HPLC) with UV-VIS detection.
  Measurements performed: Adenine Nucleotides [adenosine triphosphate (ATP), adenosine diphosphate (ADP), adenosine monophosphate (AMP), inosine monophasphate (IMP)], Guanine Nucleotides [guanosine triphosphate (GTP), guanosine diphosphate (GDP), guanosine monophosphate (GMP)].
Hypoxanthine-guanine phosphoribosyltransferase (HGPRT) activity | baseline and immediately after the intervention
  The HGPRT activity was estimated in whole blood and in erythrocytes using high-performance liquid chromatography (HPLC) with UV-VIS detection.
Nicotinamide Adenine Dinucleotide (NAD) and its metabolites | baseline and immediately after the intervention
  Nicotinamide Adenine Dinucleotide (NAD) and its metabolites were estimated in plasma using mass spectrometric procedure.
  Measurements performed: Nicotinamide Adenine Dinucleotide (NAD+), Nicotinamide (NA), 1-Methylnicotinamide (MNA), 1-methyl-2-pyridone-5-carboxamide (M2PY), 1-methyl-4-pyridone-5-carboxamide (M4PY), Nicotinamide Mononucleotide (NMN), 4-pyridone-3-carboxamide ribonucleoside (4PYR)
Total antioxidant status (TAS) | baseline
  Total antioxidant status (TAS) measurement was performed using commercially available ELISA immunoassay.
Thiobarbituric-acid-reactive substances (TBARS) | baseline
  The measurement of thiobarbituric-acid-reactive substances (TBARS) was performed using commercially available ELISA immunoassay.
Malondialdehyde (MDA) | baseline
  The measurement of malondialdehyde (MDA) was performed using commercially available ELISA immunoassay.
Polyphenols | baseline
  The measurement of polyphenols was performed using commercially available ELISA immunoassay.
Reduced glutathione (GSH) | baseline
  The measurement of reduced glutathione (GSH) was performed using commercially available ELISA immunoassay.
Glutathione peroxidase (GPx) activity | baseline
  The measurement of glutathione peroxidase (GPx) activity was performed using commercially available ELISA immunoassay.
Aminoacid profile | baseline
  The levels of 20 aminoacids were estimated in plasma using mass spectrometric procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Zieliński, Prof., Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznan University of Physical Education, Poznan, Poland

REFERENCES:
- [Derived] Pospieszna B, Kusy K, Slominska EM, Zielinski J, Ciekot-Soltysiak M. Erythrocyte nicotinamide adenine dinucleotide concentration is enhanced by systematic sports participation. BMC Sports Sci Med Rehabil. 2024 Oct 15;16(1):216. doi: 10.1186/s13102-024-00999-y. PMID 39407226